CLINICAL TRIAL: NCT04107428
Title: Somatostatin as Inflow Modulator in Adult-to-adult Living Donor Liver Transplantation: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Somatostatin in Living Donor Liver Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Collaborators: Federico II University of Naples, Department of Clinical Medicine and Surgery, Naples, Italy (Unknown); CEINGE - Biotecnologie Avanzate, Napoli, Italia (Unknown)
Responsible Party: Principal Investigator, Roberto Troisi, Principal Investigator, Clinical Professor, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C380/981/40
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: End Stage Liver DIsease; Portal Hypertension
Keywords: adult-to-adult living donor liver transplantation; small-for-size syndrome; graft hyperperfusion
MeSH Terms: conditions — End Stage Liver Disease; Hypertension, Portal | interventions — Somatostatin

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Somatostatin (Active Comparator)
  Interventions: Drug: Somatostatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Somatostatin — A bolus of 5cc of saline containing 500 mcg of somatostatin will be administered intravenously after graft reperfusion (after portal and arterial anastomosis) over a 2 minutes period, followed by a continuous infusion of 250 mcg per hour of somatostatin (infusion rate 2.5 cc/hour) for 10 days.
  Arms: Somatostatin
Drug: Placebo — A bolus of 5cc of saline will be administered intravenously after graft reperfusion (after portal and arterial anastomosis) over a 2 minutes period, followed by a continuous infusion of 2.5 cc of saline/hour for 10 days.
  Arms: Placebo

SUMMARY:
Aim of the study is to investigate the safety and the efficacy of somatostatin as liver inflow modulator in patients with end-stage liver disease (ESLD) and clinically significant portal hypertension (CSPH) undergoing Adult-to-Adult living donor liver transplantation (A2ALDLT).

DETAILED DESCRIPTION:
In liver transplantation (LT) portal hyperperfusion can severely impair graft function and survival, mainly in cases of partial LT. Perioperative somatostatin infusion has been shown to be safe, to reduce the Hepatic Vein to Portal Vein Gradients and to preserve the arterial inflow to the graft in whole liver transplantation. In partial grafts, the pharmacological action of somatostatin could reduce the graft damage due to portal hyperperfusion and arterial hypoperfusion, reducing the incidence of small-for-size syndrome and graft loss and improving the patients survival.

Objective of the study is to investigate the safety and the efficacy of somatostatin as liver inflow modulator in patients with end-stage liver disease (ESLD) and clinically significant portal hypertension (CSPH) undergoing Adult-to-Adult living donor liver transplantation (A2ALDLT).

Fifty-six patients undergoing A2ALDLT for ESLD and CSPH will be randomized double-blindly to receive somatostatin or placebo (1:1). The study drug will be administered intraoperatively as 5ml bolus (somatostatin: 500 μg), followed by a 2.5 ml/hour infusion (somatostatin: 250 μg/hour) for 10 days. Hepatic and systemic hemodynamic will be measured, along with liver function tests and clinical outcomes. The ischemia-reperfusion injury (IRI) will be analysed through histological and protein expression analysis.

The primary endpoint of the study will be the portal vein flow reduction measured at the end of liver transplant. Secondary end-points will be the reduction in the portal vein pressure, the rate of patients requiring surgical inflow modulation, the incidence of small for size syndrome, the severity of the ischemia reperfusion injury, the need for early re-transplantation (6 months), the incidence of adverse and serious adverse events, the 90-day mortality.

This randomized controlled trial could be the first to show the efficacy of somatostatin as modulator of the graft inflow in living-donor liver transplantation and potential improvement in graft and patient survival.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years old) undergoing Adult-to-Adult Living donor Liver Transplantation (LDLT) (right or left lobe)
* Indication for LDLT: End Stage Liver Disease with Portal Hypertension (HVPG ≥ 10mmHg)

Exclusion Criteria:

* Complete portal vein thrombosis (pre-operative or intraoperative diagnosis)
* Hepatopulmonary hypertension
* Adult-to-Adult Living donor liver transplantation for Fulminant hepatic failure
* Recipients of multiple solid organ transplants
* History of cardiac arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Portal venous flow changes | Day 0 - At the end of liver transplantation surgery, before skin closure
  Flow measured with transit time flow measurement system

SECONDARY OUTCOMES:
Rate of patients presenting a significant portal venous flow reduction (-20%) | Day 0 - At the end of liver transplantation surgery, before skin closure
  Flow measured with transit time flow measurement system
Rate of patients requiring surgical inflow modulation | Day 0 - At the end of liver transplantation surgery, before skin closure
Changes in hepatic artery flow | Day 0 - At the end of liver transplantation surgery, before skin closure
  Flow measured with transit time flow measurement system
Incidence of Small-for-size syndrome | 30 days
Changes in postoperative portal venous flow | Postoperative day 1, 7 and 14
  Flow measured by transabdominal ultrasound
Rates of patients requiring early re-transplantation | 6 months
Incidence of adverse and serious adverse events | 18 months
Mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Troisi, MD, PhD, Principal Investigator — King Faisal Specialist Hospital & Research Center; Dieter Broering, MD, PhD, Principal Investigator — King Faisal Specialist Hospital & Research Center

IPD SHARING:
Plan to Share IPD: No